CLINICAL TRIAL: NCT00956605
Title: A Randomized Trial of Computer-based Attention-training Systems With and Without Neurofeedback in Children With ADHD
Brief Title: A Trial of Computer-based Attention-training Systems in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: CATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Robert Bloomberg, Tufts Medical Center
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 7703
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: EEG-biofeedback; neurofeedback; computer attention training systems; ADHD; ADD; child; children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- EEG biofeedback intervention (Experimental)
  Interventions: Behavioral: Computer attention training systems for children with ADHD
- Non EEG biofeedback computerized attention training (Active Comparator)
  Interventions: Behavioral: Computer attention training systems for children with ADHD
- waitlist control (No Intervention)

INTERVENTIONS:
Behavioral: Computer attention training systems for children with ADHD — Computer attention training systems for children with ADHD, one with and one without EEG-biofeedback, were delivered via approximately 20 sessions to the participants
  Arms: EEG biofeedback intervention; Non EEG biofeedback computerized attention training

SUMMARY:
This study examines the efficacy of two computer-based training systems to teach children with ADHD to attend more effectively.

ELIGIBILITY:
Inclusion Criteria:

* child in 6th, 7th or 8th grade
* a diagnosis of ADHD (any subtype) per report of the child's physician
* academic achievement at grade level
* ability to read in English sufficiently to complete assessments and intervention protocols

Exclusion Criteria:

* coexisting diagnosis of conduct disorder, pervasive developmental disorder, or other serious mental illness (e.g., bipolar disorder, psychosis)

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2006-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Changes in ADHD symptoms as reported by caregivers and teachers were measured at enrollment pre-intervention, and then again immediately post-intervention | Assessments were administered at enrollment in May-June 2006, and then immediately post-intervention after the 3 month intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Steiner, MD, Principal Investigator — Tufts Medical Center / Tufts University
Locations (1):
- Tufts Medical Center / Tufts University, Boston, Massachusetts, United States